CLINICAL TRIAL: NCT02549807
Title: Evaluation of the Reproducibility of the Measurement by 2D Ultrasound and Sonoelastometry of the Pennation Angle and Elasticity of the Medial Gastrocnemius Muscle in Children/Adolescent/Adult Cerebral Hemiplegia After Stroke
Brief Title: Measurement by 2D Ultrasound of the Pennation Angle and Elasticity of Gastrocnemius Muscle
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1408031; 2014-A00452-45 (Other: ANSM)
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Hemiplegia
Keywords: Vascular hemiplegia; 2D ultrasound; Muscle elasticity; Pennation angle
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Children muscle elasticity measure: an ultrasound examination will be conducted on the hemiplegic leg side, while lying on his stomach and on the back. The thickness, elasticity and the angle of the medial gastrocnemius muscle pennation will be measured (muscle elasticity measure)
  Interventions: Device: Muscle elasticity measure
- Adolescent muscle elasticity measure: an ultrasound examination will be conducted on the hemiplegic leg side, while lying on his stomach and on the back. The thickness, elasticity and the angle of the medial gastrocnemius muscle pennation will be measured ((muscle elasticity measure)
  Interventions: Device: Muscle elasticity measure
- Adult muscle elasticity measure: an ultrasound examination will be conducted on the hemiplegic leg side, while lying on his stomach and on the back. The thickness, elasticity and the angle of the medial gastrocnemius muscle pennation will be measured (muscle elasticity measure)
  Interventions: Device: Muscle elasticity measure

INTERVENTIONS:
Device: Muscle elasticity measure — an ultrasound examination will be conducted on the hemiplegic leg side, while lying on his stomach and on the back. The thickness, elasticity and the angle of the medial gastrocnemius muscle pennation will be measured.

SUMMARY:
Hemiplegic adults after stroke (stroke), children and adolescents with cerebral palsy (CP) have both muscles spastic and paresis. These movement disorders are likely to cause muscle changes both structural and viscoelastic involved in the alteration of neuromotor functions such as walking. Therefore, it seems interesting to study the structure of these muscles with available imaging techniques. The medial gastrocnemius muscle presents architectural characteristics which allows easy evaluation 2D ultrasound. The literature lacks data on the reproducibility of the measurement, by 2D ultrasound, of the pennation angle and muscular thickness, particularly in children. In addition, the sonoelastometry by Supersonic ShearWave Imaging (SSI) is a new technique of ultrasound, non-invasive, dynamic, which allows the calculation of the modulus of elasticity within a muscle tissue. This allows to consider new perspectives evaluation of the viscoelastic properties of the muscle. No studies have evaluated the reproducibility of this method in adults/children/ adolescent after stroke and hemiplegia.

DETAILED DESCRIPTION:
A 1 week apart, an ultrasound examination will be conducted on the hemiplegic leg side, while lying on his stomach and on the back. The thickness, elasticity and the pennation angle of the medial gastrocnemius muscle will be measured.

ELIGIBILITY:
Inclusion Criteria:

Children

* Cerebral Paralyzed, with an infantile cerebral hemiplegia, spastic type with a level of functional independence of walking I or II of the GMFCS level.
* Having a level of spasticity in gastrocnemius muscles of the lower member plegic higher or equal to X1, V 2, on the scale of Tardieu.
* Boys aged 5 to 12 years and girls aged 5 to 11 years.

Adolescent

* Cerebral Paralyzed, with an infantile cerebral hemiplegia, spastic type with a level of functional independence of walking I or II of the GMFCS level.
* Having a level of spasticity in gastrocnemius muscles of the lower member plegic higher or equal to X1, V 2, on the scale of Tardieu.
* Boys aged 11-18 years and girls aged 10-18 years.

Adult

* Aged 18 to 75, of both sexes. - Having suffered a stroke (stroke) regardless of the date of the stroke. - Presenting hemiplegia cerebral vascular following the stroke.
* walking, with or without technical assistance or device (splint, cane ...)
* Presenting a focused plegic spasticity in the lower limb, the plantar flexors, assessed by Tardieu scale and higher than or equal to X1, V2.

Exclusion Criteria:

Children and adolescent

* Having received botulinum toxin injections in the gastrocnemius muscle in the three months preceding the assessment.
* Having received lengthening plasters in the three months preceding the assessment.
* Having benefited from therapeutic to target muscle (baclofen, a muscle relaxant ...) the beginning of the treatment would have started in the months preceding the assessment.
* Having enjoyed orthopedic surgery at the muscular structures, tendons and bone of the leg plegic.

Adult

* Presenting a concomitant muscle disease (eg myopathy, myositis ...).
* Having received injections of botulinum toxin in the gastrocnemius muscle in the three months preceding the assessment.
* Having benefited from therapeutic to target muscle (baclofen, a muscle relaxant ...) the beginning of the treatment would have started in the months preceding the assessment.
* Having enjoyed orthopedic or neurological surgery at the plegic lower limb.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hemiplegic adults/children/adolescent after stroke ,
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pennation angle | Day 1
  Pennation angle of the medial gastrocnemius muscle measuring in degrees in a sagittal section by 2D ultrasound.

SECONDARY OUTCOMES:
Muscle Elasticity | Day 1
  Measurement of elastic modulus (kPa) of anterior gastrocnemius muscles, on a sagittal section by sonoelastometry ShearWave ™.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GAUTHERON, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France